CLINICAL TRIAL: NCT03659877
Title: Identifying Physical Activity Intensity Through Accelerometry in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1617/036
Record Dates: First submitted 2017-10-25; First posted 2018-09-06 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Physical Activity; Accelerometer
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart failure patients (Experimental): Patients will be required to perform a number of physical activity tasks such as laying down, sitting and walking. During these activities, acceleration, oxygen consumption, rating of perceived exertion and heart rate will be recorded.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Participants will undertake a variety of typical daily physical activities, such as laying down, sitting, walking whilst wearing accelerometers and gas analysis equipment.

SUMMARY:
The primary objective of this study is to identify and evaluate the range of values provided by accelerometers during a variety of typical daily lifestyle activities for heart failure patients, and to relate these to the measured intensity of performing each activity in the heart failure population.

DETAILED DESCRIPTION:
The precise measurement of physical activity is now possible with advances in wearable technology, namely accelerometers. This is useful in order to properly evaluate interventions such as cardiac rehabilitation that aim to increase physical activity. One of the challenges with accelerometry is the need for raw data to be translated into meaningful behavioural units. This is addressed through a calibration study, where accelerometry data is related to oxygen consumption and cut points are derived where activity is considered light, moderate or vigorous intensity. However, calibration studies have only been done in young and healthy adults, not in the elderly or those with chronic disease such as heart failure where movements are slower and exercise capacity is reduced. This means there is a risk of underestimating the true level of physical activity in this population. Therefore the aim of this study is to run a calibration study with 18-30 heart failure patients.

Adults (aged 18 years and older) diagnosed with heart failure, with stable symptoms that are willing and able to give informed consent will be eligible for the study. Patients with contraindications to physical activity will be excluded from the study. Patients will be identified from the Royal Devon & Exeter NHS Foundation Trust and the study will be conducted in the sports science laboratory at St Luke's Campus, University of Exeter. Each patient will be required to attend a single study visit that should last approximately 3 hours in total. During the visit patients will be required to complete a number of physical activity tasks (such as lying, sitting and walking) whilst wearing various accelerometers and gas analysis equipment.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to give written informed consent to participate in study
* Adult (aged ≥18 years)
* Patients with confirmed diagnosis of heart failure
* Stable symptoms of heart failure

Exclusion Criteria:

* Patients with contraindications to exercise testing or physical activity
* Patients who are in a long term care establishment or who are unwilling or unable to travel to research site
* Patients who are unable to understand the study information.
* Patients judged to be unable to participate in the study for any other reason (e.g. diagnosis of dementia, psychiatric disorder, life-threatening comorbidity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Acceleration | Accelerometers worn for up to three hours throughout the single patient visit. Accelerometers fitted after patient signs informed consent and worn until completion of the protocol (up to 3 hours).
  acceleration (milli-g) values obtained via GENEActiv accelerometer (Activinsights, Kimbolton, UK) at multiple wear locations (both wrists, left thigh). Acceleration measured at 100Hz. Raw data reduced to one second epochs, then the average of these 1 second epochs calculated for each activity the patient completes.

SECONDARY OUTCOMES:
Oxygen consumption (VO2) | Gas analysis equipement is fitted after patient signs informed consent and worn until completion of the study protocol, up to three hours in one single patient visit.
  Breath-by-breath gas analysis. The average during the last minute of each activity the patient completes as per protocol is used.
Carbon dioxide production (VCO2) | Gas analysis equipement is fitted after patient signs informed consent and worn until completion of the study protocol, up to three hours in one single patient visit.
  Breath-by-breath gas analysis. The average during the last minute of each activity the patient completes as per protocol is used.
Respiratory Exchange Ratio (RER) | Gas analysis equipement is fitted after patient signs informed consent and worn until completion of the study protocol, up to three hours in one single patient visit.
  Breath-by-breath gas analysis. The average during the last minute of each activity the patient completes as per protocol is used.
Rating of Perceived Exertion (RPE) | This is collected throughout study completion (up to 3 hours). The patient is asked to give their RPE score during the last minute of each activity
  Borg Rating of Perceived Exertion scale (minimum score 6- maximum score 20). This is a subjective measure of how hard the patient feels they are exerting themselves.
Heart Rate | Measured throughout study completion (up to three hours). It is collected during the last minute of each activity
  Heart rate measured via pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Grace Dibben, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dibben GO, Gandhi MM, Taylor RS, Dalal HM, Metcalf B, Doherty P, Tang LH, Kelson M, Hillsdon M. Physical activity assessment by accelerometry in people with heart failure. BMC Sports Sci Med Rehabil. 2020 Aug 12;12:47. doi: 10.1186/s13102-020-00196-7. eCollection 2020. PMID 32817798